CLINICAL TRIAL: NCT07321145
Title: A Retrospective Analysis of Robot-Assisted Versus Endoscopic Breast-Conserving Surgery for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haiyan Li, chief physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-374
Record Dates: First submitted 2025-11-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic breast-conserving surgery (Active Comparator)
  Interventions: Procedure: Endoscopic breast-conserving surgery
- Robotic breast-conserving surgery (Experimental)
  Interventions: Procedure: Robotic breast-conserving surgery

INTERVENTIONS:
Procedure: Robotic breast-conserving surgery — To perform breast-conserving surgery using a robotic system, thereby validating the safety and feasibility of robotic breast-conserving surgery.
  Arms: Robotic breast-conserving surgery
Procedure: Endoscopic breast-conserving surgery — To perform breast-conserving surgery using a endoscopic system.
  Arms: Endoscopic breast-conserving surgery

SUMMARY:
Robotic surgical systems provide notable advantages including enhanced dexterity, a magnified three-dimensional high-definition view, and high-resolution imaging, thereby improving operative stability and precision. These features make robotic systems particularly suitable for procedures performed within confined operative spaces. As the breast is a solid organ without a natural cavity, robotic systems demonstrate strong adaptability for breast surgery. Robot-assisted breast-conserving surgery (RABCS) is one of the currently utilized robotic techniques in clinical breast cancer surgery. However, as robotic breast surgery remains in its early stage of development, evidence regarding the clinical outcomes of RABCS remains limited in the literature. Therefore, this study compares the surgical outcomes of endoscopic breast-conserving surgery and robot-assisted breast-conserving surgery in breast cancer patients, aiming to assess and elucidate the clinical value of RABCS.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 80 years
* Pathologically confirmed breast cancer prior to surgery
* Sufficient glandular volume with a tumor-to-breast volume ratio ≤20%
* A unifocal lesion confined to the glandular tissue
* Clear desire for breast conservation and willingness to undergo R-BCS or E-BCS
* No evidence of distant metastasis, no involvement of the skin or chest wall
* Eligibility for standard postoperative radiotherapy

Exclusion Criteria:

* The presence of diffuse suspicious lesions or microcalcifications for which wide local resection was unlikely to achieve adequate negative margins or satisfactory aesthetic outcomes
* Bilateral breast cancer or inflammatory breast cancer
* After neoadjuvant therapy, requirement for additional concurrent surgical procedures
* Inability to tolerate general anesthesia or undergo surgery
* Contraindications to radiotherapy or a history of prior chest wall irradiation, pregnancy- or lactation-associated breast cancer
* Refuse to undergo R-BCS or E-BCS

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | 1 month postoperatively

SECONDARY OUTCOMES:
Operation time | Intraoperative
Aesthetic outcomes | 3 month postoperatively
  We utilized the novel assessment tool developed by Lai et al. tailored to minimally invasive breast surgery, with specific attention to scar length, appearance, and position.
  References:
  Lai HW, Mok CW, Chang YT, Chen DR, Kuo SJ, Chen ST. Endoscopic assisted breast conserving surgery for breast cancer: Clinical outcome, learning curve, and patient reported aesthetic results from preliminary 100 procedures. Eur J Surg Oncol. 2020;46(8):1446-1455. doi:10.1016/j.ejso.2020.02.020
Blood loss | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No